CLINICAL TRIAL: NCT01587768
Title: WEUKBRE5555: IMI PROTECT (Work Package 2): The Risk of Acute Liver Injury Associated With the Use of Antibiotics
Brief Title: WEUKBRE5555: IMI PROTECT(Work Package 2): Liver Injury & Antibiotics
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 115738; WEUKBRE5559 (Other: GSK)
Record Dates: First submitted 2012-04-23; First posted 2012-04-30 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Infections, Bacterial
Keywords: Acute liver injury; antibiotics
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Time Perspective: Retrospective

GROUPS / COHORTS (3):
- Patients with a definite case of acute liver injury: The information recorded in the patients' medical record met all the criteria to be classified as idiopathic acute liver injury and the patient presents with at least with one of the following conditions (A+B or A+C):
  A - A diagnosis of liver injury (codes listed in tables 1a, 1b, 1c) with a referral to a specialist or hospital.
  Together with B - An increase of more than two times the upper limit of the normal range in alanine aminotransferase (ALT) or C - A combined increase in aspartate aminotransferase (AST), alkaline phosphatase (AP) and total bilirubin provided one of them is twice the upper limit of the respective normal range.
  Interventions: Drug: Antibiotic prescription during the study period between January 1, 2004 and December 31, 2009
- Patients with a probable case of acute liver injury: The information recorded in the patients' medical file was compatible with idiopathic acute liver injury, but not fulfilling all conditions and criteria to be defined as definite case. For example, patients identified with a READ or ICPC code for acute liver injury with a hospitalization or visit to a specialist but without complete laboratory criteria or patients identified with a READ or ICPC code for acute liver injury without a referral to a hospital/specialist, and with or without complete laboratory data.
  Interventions: Drug: Antibiotic prescription during the study period between January 1, 2004 and December 31, 2009
- Non-cases: Any potential or probable case that was excluded in one of the previous steps and those with insufficient data to determine their case status. Patients presenting normal liver function tests (LFTs), alcohol related problems, gallbladder disease, pancreatic disease, or other liver diseases with clear aetiology such as viral, alcoholic or autoimmune, or presence of other well defined pathology known to cause acute liver injury will be considered non-cases.
  Interventions: Drug: Antibiotic prescription during the study period between January 1, 2004 and December 31, 2009

INTERVENTIONS:
Drug: Antibiotic prescription during the study period between January 1, 2004 and December 31, 2009 — Antibiotics will be analysed overall, by class (tetracyclines, penicillins and betalactamics, cephalosporins, macrolides, aminoglycosides, quinolones and other antibiotics (sulphonamides & others combinations)) and individually. The antibiotics administered to patients include: cefuroxime axetil, cefuroxime sodium, ceftazidime sodium, amoxicillin, amoxicillin/ clavulanate, ampicillin, ampicillin/cloxacillin, flucloxacillin, ticarcillin, and ticarcillin/ clavulanate.

SUMMARY:
The studies described in this protocol are all performed within the framework of PROTECT (Pharmacoepidemiological Research on Outcomes of Therapeutics by a European ConsorTium) Workpackage 2 (WP2) and Workgroup 1. The primary aim of these studies is to develop, test and disseminate methodological standards for the design, conduct and analysis of Pharmacoepidemiological (PE) studies applicable to different safety issues and using different data sources. To achieve this, results from PE studies on 5 key adverse events (AEs) performed in different databases will be evaluated. Therefore, emphasis will be on the methodological aspects of the studies in this protocol and not on the clinical consequences of the association under investigation. The standards to develop will contribute to decreasing the discrepancies in results from different studies in the future and increase the usefulness and reliability of these studies for benefit-risk assessment in the EU.

We propose to assess the association between antibiotics use and idiopathic acute liver injury with different study designs (descriptive, cohort, nested case-control and case crossover) across different primary care databases and to compare the results between databases, across designs to evaluate the impact of design/database/population differences on the outcome of the studied association.

Specific aims (in each database):

1. To describe characteristics, clinical features, and risk factors for acute liver injury in patients exposed and unexposed to antibiotics.
2. To estimate the overall risk of acute liver injury associated with antibiotics exposure (users and non-users) in each database
3. To estimate the risk of acute liver injury associated with various antibiotics classes
4. To estimate the risk of acute liver injury associated with specific individual antibiotics
5. To assess the effect of dose and duration of use for specific individual antibiotics.
6. To compare the results of a case-control study with the results of a retrospective cohort study and self-controlled case series study in the different databases

The proposed studies will be collected in populations from the following databases: The General Practice Research Database [GPRD] (UK), Health Improvement Network [THIN] (UK), BIFAP [Base de datos Informatizada para estudios Farmacoepidemiologicos en Atencion Primaria] (Spain)- the Bavarian Claims Database (Germany), Mondriaan (Netherlands), and the National Databases of Denmark.

DETAILED DESCRIPTION:
Acute liver injury is one of the most important safety concerns, being the leading cause for drug withdrawal from the market on safety grounds. For most suspected hepatotoxic drugs the only existing information comes from spontaneous reports, lacking appropriate risk quantification through formal epidemiological studies. A few population-based studies examining the risk of acute and clinically relevant liver injury among users of various drugs have been published, reporting an elevated risk of liver injury in users of antibiotics. As acute liver injury is often idiosyncratic and because its diagnostic criteria used in epidemiological studies have been variable, the reported range of incidences of acute liver injury caused by antibiotics is broad. In the United Kingdom (UK), case-control studies investigating the effect of antibiotics on acute liver injury have generated odds ratios ranging from 94.8 for the combination of amoxicillin/clavulanic acid to 6.2 for tetracyclines. Age, sex, alcohol intake, concomitant medication and comorbidities have been proposed as risk factors for antibiotic induced liver injury and may have influenced the quantification of risk estimates. In the present protocol, we propose to further quantify the risk of acute liver injury associated with antibiotics in the general population using different study designs and in different primary care databases, and to compare the results to evaluate the impact of design and population differences on the outcome of the study association.

Acute liver injury or hepatotoxicity in this study implies chemical, drug driven liver damage which can be classified based on clinical presentation and laboratory features ranging from asymptomatic mild biochemical abnormalities to acute liver failure. The most common classification used for drug induced liver injury (DILI) is according to laboratory abnormalities (hepatocellular, cholestatic or mixed) and according to mechanism of toxicity (direct, immune-mediated, idiosyncratic, or mitochondrial toxicity). Being idiosyncratic in most cases, reactions often cannot be reproduced experimentally in laboratory animals. The relationship between the dose and the occurrence or severity of the reaction is not constant, and the latent period between drug exposure and sensitivity reaction is rather variable. The infrequency of DILI, though with significant impact, and complicated case ascertainment in pharmacoepidemiological studies has led to wide ranges of reported incidence rates. A recent study, using data from the GPRD database, reported crude incidence rates of liver injury caused by any type of drug ranging from 1 to 18 per 100,000 prescriptions. The Drug-Induced Liver Injury Network (DILIN), a US based collaboration between academic and health institutions to study the aetiology and prevention of DILI, found antibiotics to be the largest class of agents to cause drug-induced liver injury. UK based estimates of incidence rates of antibiotic induced liver injury range from 2.5 to 8.6 per 100,000 users.

Antibiotics are a type of antimicrobial used to treat infections and are amongst the twenty most prescribed drugs in England, with approximately 38.7 million prescriptions dispensed in 2009. The most frequently prescribed type of antibiotics is penicillins, a group of bactericidal antibiotics that interfere with bacterial cell wall synthesis. Other bactericidal antibiotics include cephalosporins and aminoglycosides. Antibiotics with bacteriostatic mechanisms of action, inhibiting the growth or proliferation of bacterial cells, include tetracyclines, macrolides, sulphonamides and quinolones. Most types of antibiotics have been associated with drug-induced liver injury.

Liver injury accounts for 10% of all adverse reactions to drugs and is the most frequent reason for withdrawal of medications from the market. This study would provide a valuable contribution to our current knowledge as drug induced liver injury is the most common cause of acute liver failure and antibiotics are the largest drug class of agents, with the highest exposure prevalence, to cause acute liver injury.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with an active or died registration status d during the study period of January 1, 2004 to December 31, 2009
* Individuals enrolled at least one year with the with the GP and having one year of computerized prescription history

Exclusion Criteria:

* Individuals with Read codes for idiopathic acute liver injury/disease, ICD-10 codes for Acute Liver injury, or CIAP codes for Idiopathic Acute Liver injury prior to start date
* Individuals with one of the following diagnoses prior to the start date: cancer, alcoholism, alcohol related problems, gallbladder disease, pancreatic disease, and other chronic liver diseases.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The primary source population will be comprised of patients of all ages with an active or died registration status during the study period of January 1, 2004 to December 31, 2009. Patients must have attained one year of enrolment with the general practioner (GP) and one year of computerized prescription history.
  From the aforementioned source population, two study cohorts will be selected.
  The first cohort will include all patients who received at least one antibiotic prescription during the study period. For this cohort, the date of first prescription of an antibiotic after meeting the eligibility criteria (entry date) defines the start of follow-up (start date), for the exposed cohort.
  The second cohort will be selected from the same source population among patients who have not received an antibiotic prescription during the study period and in the year before the entry date (date when the patient meet the eligibility criteria and enter in the study).
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2011-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Idiopathic acute liver injury | Up to six years following drug exposure
  Idiopathic acute liver injury, defined at least with one of the following conditions (A+B or A+C): A - A diagnosis of liver injury (codes listed in tables 1a, 1b, 1c) with a referral to a specialist or hospital. Together with B - An increase of more than two times the upper limit of the normal range in alanine aminotransferase (ALT) or C - A combined increase in aspartate aminotransferase (AST), alkaline phosphatase (AP) and total bilirubin provided one of them is twice the upper limit of the respective normal range.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline